CLINICAL TRIAL: NCT06618547
Title: A Study to Investigate the Effectiveness and Safety of the TENEO 317 Model 2 Excimer Laser to Treat Myopia With or Without Astigmatism by Transepithelial Photorefractive Keratectomy
Brief Title: Effectiveness and Safety of the TENEO 317 Model 2 Excimer Laser to Treat Myopia With or Without Astigmatism by Transepithelial Photorefractive Keratectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 907
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TENEO 317 Model 2 excimer laser (Experimental)
  Interventions: Device: TENEO 317 Model 2 excimer laser

INTERVENTIONS:
Device: TENEO 317 Model 2 excimer laser — TENEO 317 Model 2 excimer laser by Transepithelial Photorefractive Keratectomy

SUMMARY:
A Study to Investigate the Effectiveness and Safety of the TENEO 317 Model 2 Excimer Laser to Treat Myopia with or without Astigmatism by Transepithelial Photorefractive Keratectomy

ELIGIBILITY:
Inclusion Criteria:

1. 22 years of age or older at the time of the pre-operative examination.
2. Best distance corrected visual acuity (BCDVA) 20/25 or better in the study eye
3. Difference between manifest refractive spherical equivalent (MRSE) and the cycloplegic refraction of ≤ 0.75 D in the study eye.
4. Stable refraction (i.e., a change of ≤ 0.50 D in MRSE) for a minimum of 12 months before surgery, as verified by consecutive refractions, medical records, or prescription history.
5. Agree to discontinue contact lenses for at least two weeks (for rigid or toric lenses) or three days (for soft contact lenses) before the first refraction to establish stability and through the day of surgery.
6. A stable refraction (within ± 0.50 D) after discontinuation of contact lens(es), as determined by MRSE between two consecutive examinations at least one week apart.
7. Normal corneal topography per the investigator in the study eye.
8. Anticipated postoperative stromal thickness of at least 350 microns.
9. Ability to lie flat without difficulty.
10. Willing and able to read, understand, and sign a written informed consent form (ICF)
11. Willing and able to comply with the schedule for all post-surgery follow-up visits.
12. Pre-operative myopic refractive error with sphere component from -0.25 D to -8.00 D in each operative eye, with or without cylinder from 0.00 D to -3.00 D, based on the manifest refraction with treated MRSE of -0.25 D to -9.50 D.

Exclusion Criteria:

1. Acute or chronic disease or illness that would increase operative risk or confound the results of the study (e.g., dry eye, cataract, immuno-compromise, rheumatoid arthritis, clinically significant atopic disease, acne rosacea, autoimmune disease, endocrine disorders, lupus, systemic connective tissue disease, diabetes, or severe atopic disease).
2. Use of medications that may increase risk to the subject or may confound the outcome of the study, including those known to affect wound healing (e.g., systemic corticosteroids, antimetabolites)
3. Ocular conditions that may predispose the subject to future complications, including but not limited to:

   1. Evidence or history of retinal vascular disease
   2. History or evidence of active corneal disease or infection (e.g., recurrent corneal erosion syndrome, herpes simplex or herpes zoster keratitis) in either eye.
   3. History of or evidence of glaucoma or glaucoma suspect (e.g., IOP > 21 mmHg).
4. Previous intraocular or corneal surgery in an eye considered for eligibility that might confound the study's outcome or increase the subject's risk.
5. An increased risk for developing strabismus post-treatment or an ocular muscle disorder (e.g., strabismus or nystagmus) affecting fixation.
6. Known sensitivity to any study medications (e.g., used during TransEpi PRK procedure and postoperative care).
7. Central corneal scars affecting visual acuity.
8. Presence of keratoconus, subclinical or forme fruste keratoconus, corneal dystrophy, or other corneal irregularity (e.g., irregular astigmatism).
9. Presence of visually significant or progressive cataract in an eye considered for eligibility.
10. Actively taking medications contraindicated with TransEpi PRK, such as isotretinoin (Accutane®) or amiodarone hydrochloride (Cordarone®).
11. Cardiac pacemaker, implanted defibrillator, or another implanted electronic device.
12. Pregnant, lactating, or subjects who plan to become pregnant during the study.
13. Participation in any other clinical trial within 30 days of screening or during this clinical trial.14. Subjects for whom the pre-operative assessment of the cornea/ eyes indicates that one or both eyes are not suitable candidates for treatment based upon the investigator's medical judgment.

15. Treated eye with mesopic pupil size > 7.0 mm.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Maintenance of BCDVA - | through study completion, an average of 1 year
  lines lost <5% of eyes with a loss of >2 lines of BCDVA at the stability visit
Maintenance of BCDVA - | through study completion, an average of 1 year
  preservation 20/40 <1% of eyes with a BCDVA of 20/20 or better preoperatively that have a BCDVA worse than 20/40 at the stability visit
Induced manifest refractive astigmatism | through study completion, an average of 1 year
  <5% of eyes with induced manifest refractive astigmatism greater >2 diopters at the stability visit
Induced manifest refractive astigmatism | through study completion, an average of 1 year
  < 1% of eyes with serious adverse events by type of event observed through the final study visit.

IPD SHARING:
Plan to Share IPD: No